CLINICAL TRIAL: NCT05786183
Title: Diagnostic Accuracy of a Rapid Technique for the Detection of Intestinal Anti-transglutaminase Antibodies to Enable a Real Time Diagnosis of Celiac Disease
Brief Title: Rapid Technique for the Detection of Intestinal Anti-transglutaminase Antibodies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 34/20
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Coeliac Disease
Keywords: intestinal antibodies; Rapid test; Coeliac disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intestinal Celiac Disease (CD)-antibodies have been described as the best marker to reveal progression toward villous atrophy and could become the diagnostic marker to make prompt diagnosis in the wide clinical spectrum of CD reducing the delay in diagnosis and treatment. The introduction of either anti-endomysial antibodies (EMA) assay or rapid anti-Transglutaminase 2 (TG2) test on supernatant of mechanically lysed biopsy samples in the clinical practice would improve the diagnosis of CD, especially in clinically challenging scenarios. The availability of an accurate test for identifying intestinal CD-antibodies that do not need the culture of intestinal biopsy is less expensive, less time consuming and easier to perform would facilitate the implementation of such technology outside research laboratories, and enable the diagnosis of CD at the end of Gastrointestinal Endoscopy (GIE).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective esophagogastroduodenoscopy (EGD) for suspected CD, eosinophilic esophagitis, autoimmune enteropathy, inflammatory bowel disease, gastritis, gastric or duodenal ulcer, gastroesophageal reflux disease.

Exclusion Criteria:

* Bleeding disorders
* Patients fulfilling the new ESPGHAN Guidelines for diagnosing CD (version 2020), for a serology based CD diagnosis
* Subjects in whom intestinal biopsies are not indicated as part of the diagnostic process.

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects included in the study will be children and young adults, between 1 to 22 years of age, referred to the Gastroenterology Unit for elective GIE
Sampling Method: Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of EMA assay detected on supernatant of mechanically lysed intestinal biopsy specimens | At the time of endoscopic examination
  Sensitivity and specificity of EMA assay detected on mechanically lysed intestinal biopsies compared to the reference standard (serology + histopathology)
Diagnostic accuracy of rapid anti-TG2 test detected on supernatant of mechanically lysed intestinal biopsy specimens | At the time of endoscopic examination
  Sensitivity and specificity of rapid anti-TG2 test detected on mechanically lysed intestinal biopsies compared to the reference standard (serology + histopathology)

SECONDARY OUTCOMES:
Concordance of EMA assay and rapid anti-TG2 test on supernatant of mechanically lysed intestinal biopsy specimens with Culture-EMA results | At the time of endoscopic examination

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided